CLINICAL TRIAL: NCT07128472
Title: Evaluation of IL 12B Genetic Polymorphism (rs3213094) in Patient With Psoriasis and Psoriatic Arthritis in Response to Humira
Brief Title: Evaluation of IL 12B Genetic Polymorphism (rs3213094)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Alaa Ahmed Saad Ali Aweida, Resident at Dermatology , venereology and andrology, Faculty of medicine, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SVU-MED-DVA021-4
Record Dates: First submitted 2025-08-13; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients Group (Active Comparator): About 20 patients with psoriasis and psoriatic arthritis.
  Interventions: Drug: Humira
- Healthy Group (Active Comparator): About 20 healthy control group.
  Interventions: Drug: Humira

INTERVENTIONS:
Drug: Humira — Assess the response of psoriasis and psoriatic arthritis to Humira and also Assessing the pharmacogenetic association between IL 12B genetic polymorphism (rs3213094) in psoriatic and psoriatic arthritis patients taking Humira.
  Other Names: IL 12B genetic polymorphism (rs3213094)

SUMMARY:
Psoriasis is a skin disorder that is chronic proliferative and inflammatory in nature. Extensor surfaces, scalp, and lumbosacral area are covered in erythematous plaques with silvery scales. The disease can also impair the eyes and joints. It has no cure. Because of their low quality of life, many psoriasis patients experience depression. In addition to the cutaneous manifestations, it is associated with an increased risk of psoriatic arthritis, depression and cardiovascular disease.

DETAILED DESCRIPTION:
Psoriasis is known to be affecting 3% to 4% of the general population worldwide. While the prevalence of psoriasis in Egypt ranges 0.19-3% Psoriatic arthritis (PsA) most commonly develops in 20-30% of psoriatic patients with preceding psoriasis or develops concomitantly with psoriasis, and it manifests all features of arthritis, including enthesitis.

The pathogenesis of psoriasis is multifactorial, involving a complex interplay between genetic predisposition, immune system dysregulation, and environmental triggers. Central to the disease process is the activation of T-cells, particularly Th1, Th17, and Th22 subsets, which release pro-inflammatory cytokines such as tumor necrosis factor-alpha (TNF-α), interleukin-17 (IL-17), and interleukin-22 (IL-22)

. These cytokines drive the abnormal growth and differentiation of keratinocytes and induce the inflammatory cascade that results in the characteristic skin lesions. Genetic factors, including polymorphisms in genes related to the immune system, such as HLA-Cw6.Additionally, environmental factors like infections, stress, and trauma (Koebner phenomenon) can exacerbate or trigger the onset of the disease.

The Psoriasis Area and Severity Index (PASI) is a widely used tool for assessing the severity of psoriasis and evaluating treatment efficacy. It combines the extent of skin involvement and the degree of erythema, scaling, and thickness across four body regions: the head, upper limbs, trunk, and lower limbs. Each region is assigned a score for surface area involvement (0-6) and for each symptom (0-4), which are then combined to yield an overall PASI score ranging from 0 to 72. Higher scores indicate more severe disease. Typically, a PASI score below 10 suggests mild psoriasis, while scores between 10 and 20 indicate moderate severity, and scores above 20 reflect severe psoriasis. PASI serves as a critical endpoint to gauge disease burden.

Interleukin-12B (IL12B) encodes the p40 subunit shared by both IL-12 and IL-23, cytokines that are pivotal in the differentiation of naive T-cells into Th1 and Th17 cells, respectively. The IL-12/IL-23 axis is well-established in contributing to the immune pathology seen in psoriasis. Genetic studies have shown that polymorphisms within the IL12B gene are associated with an increased risk of psoriasis.

Single nucleotide polymorphisms (SNPs) are the most common type of genetic variation in humans. SNP rs3213094, located within the IL12B gene, has been identified as a potentially significant variant that could alter the expression or function of the cytokines involved in immune responses. Previous studies have suggested that SNP rs3213094 within the IL12B gene is associated with psoriasis, although the strength of this association varies across different populations.

Humira (adalimumab) is a monoclonal antibody targeting TNF-α, widely used for treating moderate-to-severe psoriasis and PsA. It works by neutralizing the activity of TNF-α, thereby reducing inflammation, decreasing keratinocyte proliferation, and alleviating joint symptoms. However, individual responses to Humira can vary significantly, with some patients experiencing limited or no therapeutic benefits

ELIGIBILITY:
Inclusion Criteria:

- Patients having psoriasis diagnosed clinically for at least 6 months and who have a severity grade of severe, defined as a Psoriasis Area and Severity Index (PASI) score greater than 10, and involvement of greater than 10% of the body surface area (BSA) with psoriatic arthritis.

Exclusion Criteria:

* Patients with other autoimmune or inflammatory conditions (e.g., rheumatoid arthritis, lupus).
* Pregnancy and lactation.
* Patients currently undergoing any treatment other than Humira.
* Patients with known genetic disorders affect immune system function.
* Patients were undergoing any treatment other than Humira in the last 6 months.
* Patients with active infections, including tuberculosis or chronic viral infections (e.g., hepatitis B or C, HIV).
* Patients with contraindication to Humira.
* Renal &Vascular diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Treatment of Psoriasis and Psoriatic Arthritis | 3 Months
  Treatment the patients whom suffering from Psoriasis and Psoriatic arthritis and Assessment of clinical improvement to Humira therapy according to: PASI score into PASI 50: means 50% reduction in PASI score - an acceptable measure of efficacy for secondary endpoints in psoriasis clinical trials PASI 75: means 75% reduction in PASI score - standard efficacy measure used in most psoriasis clinical studies1 PASI 90: means 90% reduction in PASI score (almost clear skin) PASI 100: means Completely clear skin.

SECONDARY OUTCOMES:
Evaluate the effect of treatment with Humira | 3 Months
  Evaluate the effect of treatment with Humira therapy on the level of serum IL12B genetic polymorphism (rs3213094) on the Participants whom suffering from Psoriasis and Psoriatic arthritis.

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa Adam Ali El Taieb, Professor, Study Chair — Dermatology, Venereology and Andrology. Faculty of Medicine,Qena University; Eisa Mohammed Hegazy, Professor, Study Director — Dermatology, Venereology and Andrology. Qena Faculty of Medicine,South Valley University; Mohamed Hosny Hassan, Professor, Principal Investigator — Medical Biochemistry Department,Qena Faculty of Medicine,south valley university
Locations (1):
- Qina University hospital, South Valley University Hospital, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Undecided